CLINICAL TRIAL: NCT05641428
Title: A Phase II Non-inferiority Study Comparing Point-of-care Produced CAR T-cell to Commercial CAR T-cells in Patients with Relapsed/refractory Non-Hodgkin Lymphoma
Brief Title: Comparison of Point-of-care Produced CAR T-cell with Commercial CAR T-cells in Patients with R/R LBCL
Acronym: HOVON161
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HO161 CAR T; 2021-000937-15 (EudraCT Number)
Record Dates: First submitted 2022-10-11; First posted 2022-12-07 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: NHL; DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (ARI-0001) (Experimental): Infusion with Point of Care CAR T-cells
  Interventions: Drug: ARI-0001
- Arm B (Axi-cel) (Active Comparator): Infusion with Standard of Care CAR T-cells
  Interventions: Drug: Axi-cel

INTERVENTIONS:
Drug: ARI-0001 — Infusion with a single target dose of 2.0 x 10^6 Point of Care CAR T-cells/kg BW (range 1 -2.0x 10^6 CAR T-cells /kg BW).
  Arms: Arm A (ARI-0001)
Drug: Axi-cel — Infusion with a single target dose of 2.0 x 10^6 Standard of Care CAR T-cells/kg BW (range 1 -2.0x 10^6 CAR T-cells /kg BW).
  Arms: Arm B (Axi-cel)

SUMMARY:
A phase II, multi-center study to compare the feasibility, and clinical efficacy of local manufacturing of CD19-directed CAR T-cells (ARI-0001 CAR T-cells) with commercial produced CAR T-cells (for example axicabtagene ciloleucel, a CD19 targeting commercially available CAR T-cell) in patients with relapsed or refractory (R/R) DLBCL.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) T-cell therapy is an innovative form of adoptive cell therapy that has proven its efficacy in the treatment of various hematological malignancies, including B-cell non-Hodgkin lymphoma (NHL) and B-cell acute lymphoblastic leukemia (ALL). CD19 has been the most studied target antigen for CAR T-cell immunotherapy. Anti-CD19 CAR T-cell therapy has shown durable responses in patients with different B-NHLs, including Diffuse Large B-cell Lymphoma (DLBCL).

Unfortunately, up to 50-60% of the patients do not respond to CD19-directed CAR T-cell therapy or relapse. There are several shortcomings of current CD19-directed CAR T-cell therapy, that are likely responsible for therapy failure, namely: i) Due to centralized production at commercial sites, the production is time consuming (about 4 weeks), meaning that patients with rapidly progressive lymphoma may not reach the moment of the infusion of the anti-CD19 CAR T-cells. ii) Furthermore, for the current production processes, the autologous T-cells need to be cryopreserved for shipment from the hospital to the production sites and vice versa. This (double) cryopreservation process can decrease the quality of the CAR T-cells. This trial aims to address these shortcomings and will study the feasibility, and clinical efficacy of local manufacturing of CD19-directed CAR T-cells (ARI-0001 CAR T-cells), in a completely closed system using the CliniMACS Prodigy device. This study will compare the clinical efficacy of locally produced CAR T-cells to commercial produced CAR T-cells (for example axicabtagene ciloleucel, a CD19 targeting commercially available CAR T-cell) in patients with relapsed or refractory (R/R) DLBCL.

This in-house (point-of-care) production process of ARI-0001 will take approximately 7-12 days and thus will generate CAR T-cells "faster" which will be infused in the patient without cryopreservation ("fresh", of note, a back-up cryopreserved product will also be manufactured). Furthermore, the point-of-care production process can be replicated in academic institutions with the appropriate cellular manufacturing facilities. If successful, this study will show feasibility of local production of CAR T-cell therapy, improving their rapid accessibility and quality.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLBCL and associated subtypes, defined by WHO 2016 classification: DLBCL not otherwise specified (NOS), High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (DHL/THL) and FL3B, T-cell/histocyte rich B-cell lymphoma, Primary mediastinal B-cell lymphoma, transformed lymphoma (transformed follicular) and R/R after at least 2 lines of systemic therapy
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG)/WHO performance status 0-2
* Secondary central nervous system (CNS) involvement is allowed however, then he/she must have

  * No signs or symptoms of CNS involvement that would hamper adequate ICANS assessment
* Estimated life expectancy of >3 months other than primary disease
* Patients of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen
* Signed and dated informed consent before conduct of any trial-specific procedure
* Patient is capable of giving informed consent

Exclusion Criteria:

* Absolute neutrophil count (ANC) <1.0x10^9/L
* Platelet count <50x10^9/L
* Absolute lymphocyte count <0.1x10^9/L
* Primary CNS lymphoma
* Known history of infection with hepatitis C or B virus unless treated and confirmed to be polymerase chain reaction (PCR) negative
* Active HIV infection with detectable viral load or CD4 T-cell count below 0.20x10^9/L
* Known history or presence of seizure activities or on active anti- seizure medications within the previous 12 months
* Known history of CVA within prior 12 months
* Unstable neurological deficits
* Known history or presence of autoimmune CNS disease, such as multiple sclerosis, optic neuritis or other immunologic or inflammatory disease
* Active systemic autoimmune disease for which immunosupressive therapy is required
* Presence of CNS disease that, in the judgment of the investigator, may impair the ability to evaluate neurotoxicity, baseline dementia that would interfere with therapy or monitoring, determined using mini-mental status exam at baseline
* Active systemic fungal, viral or bacterial infection
* Clinical heart failure with New York Heart Association class ≥2 (appendix F) or Left Ventricular Ejection Fraction (LVEF) <40%
* Resting oxygen saturation <92% on room air
* Liver dysfunction as indicated by total bilirubin, AST and/or ALT >5 x institutional ULN, unless directly attributable to the lymphoma or Gilbert disease
* GFR <40 mL/min calculated according to the modified formula of Cockcroft and Gault or by direct urine collection
* Pregnant or breast-feeding woman
* Active other malignancy requiring treatment
* Medical condition requiring prolonged use of systemic immunosuppressives with exception of prednisolone <10 mg/day
* History of severe immediate hypersensitivity reaction against any drug or its Ingredients/impurities that is scheduled to be given during trial participation e.g. as part of the mandatory lymphodepletion protocol, premedication for infusion, or rescue medication/salvage therapies for treatment related toxicities
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) from date of IMP infusion (if applicable) | Approximately up to 60 months following first patient IMP infusion
  PFS from date of IMP infusion is defined as the time from IMP infusion, until progression, relapse or death from any cause, whichever comes first. PFS reflects tumor growth and, therefore, occurs prior to the endpoint of OS. Progression is defined as the first date of documentation of a new lesion or enlargement of a previous lesion, or the date of the scheduled clinic visit immediately after radiologic assessment has been completed. If there is missing information, censoring of the data may be defined as the last date at which progression status was adequately assessed.

SECONDARY OUTCOMES:
Progression-free survival (PFS) from date of randomization | Approximately up to 60 months following first patient enrollment
  PFS from date of randomization is defined as the time from enrollment, until progression, relapse or death from any cause, whichever comes first. PFS reflects tumor growth and, therefore, occurs prior to the endpoint of OS. Progression is defined as the first date of documentation of a new lesion or enlargement of a previous lesion, or the date of the scheduled clinic visit immediately after radiologic assessment has been completed. If there is missing information, censoring of the data may be defined as the last date at which progression status was adequately assessed.
Safety and toxicity assessment per AE reporting | Approximately up to 60 months following first patient IMP infusion
  Safety and toxicity assessment of ARI-0001 CAR T-cells and Axi-cel per AE reporting classified according to CTCAE Version 5 and CRS and ICANS classified according to the ASTCT criteria. The number and proportion of patients in the specific safety population with CTCAE grade 2, 3 or 4 (incl. grade 5) will be tabulated by randomization arm. Per site, the maximum observed grade per cycle within a patient will be used.
Overall Response Rate (ORR) | At 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells
  ORR is the sum of complete response (CR) and partial response (PR), as well as CR, PR, SD and PD/relapse at 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells.
Expansion of CAR T-cells | Approximately up to 60 months following first patient IMP infusion
  Expansion of CAR T-cells will be assessed in both treatment arms. The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
Phenotype of CAR T-cells | Approximately up to 60 months following first patient IMP infusion
  Phenotype of CAR T-cells will be assessed in both treatment arms. The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
Persistence of CAR T-cells | Approximately up to 60 months following first patient IMP infusion
  Persistence of CAR T-cells will be assessed in both treatment arms. The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
Best Overall Response (BOR) | 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells
  BOR is the best response recorded from randomization until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started) or start treatment in follow up, whichever occurs first. The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. It will be analyzed at 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells.
Duration Of Response (DOR) | Approximately up to 60 months following first patient IMP infusion
  DOR is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until time of the last assessment of response before the first date that recurrent or progressive disease is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started). New treatment in follow up or death without previous recurrent or progressive disease will be considered as competing risks.
Overall Survival (OS) | Approximately up to 60 months following first patient IMP infusion
  OS is defined as the time from date of enrollment or from IMP infusion to the date of death from any cause (2 separate endpoints). Patients still alive will be censored at the date of last contact.
Patient Reported Outcome/Quality of Life (PRO/QOL) EuroQol- 5 Dimension (EQ-5D) | At 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells
  PRO/QOL will be assessed using the EQ-5D. Questionnaire will be completed by the subject, after registration and prior to leukapheresis, at 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells.
  The EQ-5D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Patient Reported Outcome/Quality of Life (PRO/QOL) Functional Assessment of Cancer Treatment-Lymphoma (FACT-Lym) | At 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells
  PRO/QOL will be assessed using FACT-Lym. Questionnaire will be completed by the subject, after registration and prior to leukapheresis, at 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells.
  The FACT-Lym (Functional Assessment of Cancer Therapy - Lymphoma) comprises Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Lymphoma Subscale using a 5 point Likert-type scale.
Patient Reported Outcome/Quality of Life (PRO/QOL) Quality of Life Questionnaire (QLQ-C30) | At 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells
  PRO/QOL will be assessed using QLQ-C30. Questionnaire will be completed by the subject, after registration and prior to leukapheresis, at 4 weeks, 12 weeks, 6, 12 and 24 months after infusion of CAR T-cells.
  The QLQ-C30 is a Quality of Life questionnaire designed to measure cancer patients' physical, psychological and social functions, composed of both multi-item scales and single-item measures.
PoC CAR T-cell production characteristics (e.g. number of viable T-cells) | Approximately up to 60 months following first patient with PoC IMP infusion
  PoC CAR T-cell production characteristics (e.g. number of viable T-cells), including the functional characteristics (e.g. potency tests) between the different production sites. The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
PoC CAR T-cell production characteristics (e.g. transduction efficiency) | Approximately up to 60 months following first patient with PoC IMP infusion
  PoC CAR T-cell production characteristics (e.g. transduction efficiency), including the functional characteristics (e.g. potency tests) between the different production sites. The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
PoC CAR T-cell production characteristics (e.g. T-cell subsets (activated T-cells, memory T-cells)) | Approximately up to 60 months following first patient with PoC IMP infusion
  PoC CAR T-cell production characteristics (e.g. T-cell subsets (activated T-cells, memory T-cells)), including the functional characteristics (e.g. potency tests) between the different production sites. The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
The association of the functional characteristics (e.g. potency tests) of the CAR T-cell products (ARI-0001 CAR T-cells) with CAR T-cell expansion. | Approximately up to 60 months following first patient with PoC IMP infusion
  The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
The association of the functional characteristics (e.g. potency tests) of the CAR T-cell products (ARI-0001 CAR T-cells) with CAR T-cell persistence. | Approximately up to 60 months following first patient with PoC IMP infusion
  The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
The association of the functional characteristics (e.g. potency tests) of the CAR T-cell products (ARI-0001 CAR T-cells) with CAR T-cell adverse events. | Approximately up to 60 months following first patient with PoC IMP infusion
  The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
The association of the functional characteristics (e.g. potency tests) of the CAR T-cell products (ARI-0001 CAR T-cells) with CAR T-cell response rates. | Approximately up to 60 months following first patient with PoC IMP infusion
  The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
The association of the functional characteristics (e.g. potency tests) of the CAR T-cell products (ARI-0001 CAR T-cells) with CAR T-cell progression free survival. | Approximately up to 60 months following first patient with PoC IMP infusion
  The central lab will collect these data, but the vast majority will not be entered in the ALEA database, and will only be analyzed by the central lab. Further details and analyses will be described in a separate SAP, which will be written by those involved in that specific analysis.
Proportion of successful batches (in percentage) between the different production sites. | Approximately up to 60 months following first patient with PoC IMP infusion
Number of days between leukapheresis and infusion of CAR T-cells (vein-to-vein time) | Approximately up to 60 months following first patient IMP infusion

CONTACTS AND LOCATIONS:
Overall Officials: T. (Tom) van Meerten, Principal Investigator — UMCG / HOVON
Locations (7):
- Netherlands (7):
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Groningen-UMCG, Groningen
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Utrecht-UMCUTRECHT, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.hovon.nl